CLINICAL TRIAL: NCT02073162
Title: REstrictive Versus LIbEral Fluid Therapy in Major Abdominal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 13-1287
Record Dates: First submitted 2014-02-21; First posted 2014-02-27 (Estimated); Results first posted 2019-10-31 (Actual); Last update posted 2019-10-31 (Actual); Status verified 2019-10

CONDITIONS: Major Abdominal Surgery

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Liberal group (Active Comparator): At induction-Hartmanns 10 ml/kg During surgery-Hartmanns 8 ml/kg/h After surgery-IV fluids ≥1.5 ml/kg/h Continue IV fluids ≥24hrs
  Interventions: Procedure: Major Abdominal Surgery
- Restrictive group (Experimental): At induction-Hartmanns ≤5 ml/kg During surgery-Hartmanns 5 ml/kg/h After surgery-IV fluids, ≤0.8 ml/kg/h Cease IV fluids ASAP,aim for early oral fluids
  Interventions: Procedure: Major Abdominal Surgery

INTERVENTIONS:
Procedure: Major Abdominal Surgery — •All types of open or lap-assisted abdominal or pelvic surgery with an expected duration of at least 2 hours, and an expected hospital stay of at least 3 days (for example, oesophagectomy, gastrectomy, pancreatectomy, colectomy, aortic or aorto-femoral vascular surgery, nephrectomy, cystectomy, open prostatectomy, radical hysterectomy, and abdominal incisional hernia repair)

SUMMARY:
Physicians differ in their approaches to surgical fluid therapy, with some preferring higher volumes and others lower volumes. Each approach has potential advantages and disadvantages. Currently, there is no compelling evidence that one approach is better than the other. This study tests whether giving a volume on the low end of the usual amount ("restrictive management") has a different rate of complications compared to a volume on the high end of the usual amount ("liberal management"). This study will compare liberal and restrictive fluid management to determine their effects on major complications after abdominal surgery.

Those who take part in the study will be visited five times before and after surgery in the hospital. Once discharged from the hospital, participants will be called 4 times on the telephone.

Preadmission Clinic/Preoperative Visit

* Sign the consent document
* Have blood drawn for standard preoperative tests (standard of care)
* Have an electrocardiogram (standard of care)
* Complete a questionnaire on disability (research)

Day of Surgery

* Have blood drawn if not already done during the first visit (standard of care)
* Have an electrocardiogram if not already done during the first visit (standard of care)
* Be randomly assigned to either restrictive or liberal fluid management (research)

Post-op Day 1

* Have an electrocardiogram done (research)
* Have blood drawn for standard tests (standard of care)
* Have a wound inspection, if there is a change of dressing (standard of care)
* Complete a questionnaire about your recovery (research)

Post-op Day 3

* Have blood drawn for standard tests (standard of care) and c-reactive protein, which can indicate infection (for research).
* Have a wound inspection, if there is a change of dressing (standard of care)
* Complete a questionnaire about your recovery (research)

Day of Discharge

* Have a wound inspection, if there is a change of dressing (standard of care)

  30-Day Follow-up Phone Call
* Complete a questionnaire about your recovery (research)
* Complete a questionnaire about disability (research)

  3 Month, 6-Month, and 12-Month Follow-up Phone Calls
* Complete a questionnaire about disability (research)

ELIGIBILITY:
Inclusion Criteria:

* adults (≥18 years) undergoing elective major surgery and providing informed consent
* all types of open or lap-assisted abdominal or pelvic surgery with an expected duration of at least 2 hours, and an expected hospital stay of at least 3 days (for example, oesophagectomy, gastrectomy, pancreatectomy, colectomy, aortic or aorto-femoral vascular surgery, nephrectomy, cystectomy, open prostatectomy, radical hysterectomy, and abdominal incisional hernia repair)
* at increased risk of postoperative complications, defined as at least one of the following criteria:
* age ≥70 years
* known or documented history of coronary artery disease
* known or documented history of heart failure
* diabetes currently treated with an oral hypoglycaemic agent and/or insulin
* preoperative serum creatinine >200 μmol/L (>2.8 mg/dl)
* morbid obesity (BMI ≥35 kg/m2)
* preoperative serum albumin <30 g/L
* anaerobic threshold (if done) <12 mL/kg/min
* or two or more of the following risk factors:
* ASA 3 or 4
* chronic respiratory disease
* obesity (BMI 30-35 kg/m2)
* aortic or peripheral vascular disease
* preoperative haemoglobin <100 g/L
* preoperative serum creatinine 150-199 μmol/L (>1.7 mg/dl)
* anaerobic threshold (if done) 12-14 mL/kg/min

Exclusion Criteria:

* urgent or time-critical surgery
* ASA physical status 5 - such patients are not expected to survive with or without surgery, and their underlying illness is expected to have an overwhelming effect on outcome (irrespective of fluid therapy)
* chronic renal failure requiring dialysis
* pulmonary or cardiac surgery - different pathophysiology, and thoracic surgery typically have strict fluid restrictions
* liver resection - most units have strict fluid/CVP limits in place and won't allow randomisation
* minor or intermediate surgery, such as laparoscopic cholecystectomy, transurethral resection of the prostate, inguinal hernia repair, splenectomy, closure of colostomy - each of these are typically "minor" surgery with minimal IV fluid requirements, generally low rates of complications and mostly very good survival.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3000 (Actual)
Dates: Start 2014-02; Primary Completion 2016-09 (Actual); Study Completion 2018-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Kurz, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Liberal Group | Restrictive Group
Started | 1499 | 1501
Completed | 1493 | 1490
Not Completed | 6 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Liberal Group | Restrictive Group | Total
Number analyzed (Participants) | 1493 | 1490 | 2983
Age, Continuous [Mean (Standard Deviation); unit: years] | 66 (13) | 66 (13) | 66 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 710 | 719 | 1429
  Male | 783 | 771 | 1554
Region of Enrollment [Count of Participants; unit: Participants]
  Australia | 841 | 836 | 1677
  Canada | 247 | 250 | 497
  United Kingdom | 134 | 141 | 275
  Hong Kong | 116 | 111 | 227
  United States | 75 | 74 | 149
  New Zealand | 48 | 46 | 94
  Italy | 32 | 32 | 64
Body Weight [Median (Inter-Quartile Range); unit: kg] | 83 [69 to 102] | 84 [68 to 102] | 83 [68 to 102]
ASA Physical Status Classification [Count of Participants; unit: Participants] — ASA I: A normal healthy patient ASA II: A patient with mild systemic disease ASA III: A patient with severe systemic disease ASA IV: A patient with severe systemic disease that is a constant threat to life
  Participants
    ASA I | 21 | 25 | 46
    ASA II | 540 | 542 | 1082
    ASA III | 868 | 849 | 1717
    ASA IV | 64 | 74 | 138
Median preoperative WHODAS score [Median (Inter-Quartile Range); unit: units on a scale] — World Health Organization Disability Assessment Schedule (12 item) estimates the amount of disability. Each of the item in the questionnaire scores from 0 (No difficulty) to 4 (Extreme Difficulty or Cannot Do). The total score summed over the 12 items for the whole questionnaire ranges from 0 to 48, with the score of 24 or greater indicating at least moderate disability.
  units on a scale | 15 [13 to 21] | 15 [13 to 21] | 15 [13 to 21]
Hypertension [Count of Participants; unit: Participants] | 908 | 899 | 1807
Coronary artery disease [Count of Participants; unit: Participants] | 250 | 212 | 462
Heart failure [Count of Participants; unit: Participants] | 47 | 57 | 104
Previous myocardial infarction [Count of Participants; unit: Participants] | 146 | 122 | 268
Peripheral vascular disease [Count of Participants; unit: Participants] | 92 | 95 | 187
Current smoker [Count of Participants; unit: Participants] | 204 | 194 | 398
History of stroke or TIA [Count of Participants; unit: Participants] | 115 | 105 | 220
Chronic obstructive pulmonary disease [Count of Participants; unit: Participants] | 254 | 244 | 498
Moderate or severe renal disease [Count of Participants; unit: Participants] | 108 | 101 | 209
Neuraxial block [Count of Participants; unit: Participants] | 358 | 409 | 767
Invasive blood-pressure monitoring [Count of Participants; unit: Participants] | 1080 | 1070 | 2150
CVP monitoring [Count of Participants; unit: Participants] | 272 | 276 | 548
Type of Surgery [Count of Participants; unit: Participants]
  Esophageal or gastric | 257 | 286 | 543
  Hepatobiliary | 139 | 133 | 272
  Colorectal | 651 | 646 | 1297
  Urologic or renal | 223 | 220 | 443
  Gynecologic | 139 | 135 | 274
  Other | 84 | 70 | 154
Surgical method [Count of Participants; unit: Participants]
  Open | 788 | 818 | 1606
  Laparoscopic | 463 | 458 | 921
  Laparoscopic-assisted | 242 | 214 | 456
Duration of Surgery [Median (Inter-Quartile Range); unit: hr] | 3.3 [2.5 to 4.5] | 3.3 [2.4 to 4.6] | 3.3 [2.4 to 4.6]
Planned postoperative care in HDU or ICU [Count of Participants; unit: Participants] | 418 | 416 | 834

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Disability-free Survival
Description: Disability was defined as a persistent impairment in health status (lasting ≥6 months), as measured by a score of at least 24 points on the WHODAS questionnaire, which reflects a disability level of at least 25% (the threshold point between "disabled" and "not disabled").
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Liberal Group | Restrictive Group
Number analyzed (Participants) | 1493 | 1490
Participants | 1232 | 1223

2. Secondary Outcome: Number of Participants With Acute Kidney Injury
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Liberal Group | Restrictive Group
Number analyzed (Participants) | 1493 | 1490
Participants | 72 | 124

3. Secondary Outcome: Number of Participants With a Composite of Mortality or Major Septic Complications
Time Frame: 30-day
Measure: Count of Participants; unit: Participants
Arm/Group | Liberal Group | Restrictive Group
Number analyzed (Participants) | 1493 | 1490
Participants | 195 | 323

4. Secondary Outcome: Number of Participants With Surgical-site Infection
Time Frame: Indexed hospital stay
Measure: Count of Participants; unit: Participants
Arm/Group | Liberal Group | Restrictive Group
Number analyzed (Participants) | 1493 | 1490
Participants | 202 | 245

5. Secondary Outcome: Number of Participants With Sepsis
Time Frame: Indexed hospital stay
Measure: Count of Participants; unit: Participants
Arm/Group | Liberal Group | Restrictive Group
Number analyzed (Participants) | 1493 | 1490
Participants | 129 | 157

6. Secondary Outcome: Number of Participants With Anastomotic Leak
Time Frame: Indexed hospital stay
Measure: Count of Participants; unit: Participants
Arm/Group | Liberal Group | Restrictive Group
Number analyzed (Participants) | 1493 | 1490
Participants | 35 | 49

7. Secondary Outcome: Number of Participants With Pneumonia
Time Frame: Indexed hospital stay
Measure: Count of Participants; unit: Participants
Arm/Group | Liberal Group | Restrictive Group
Number analyzed (Participants) | 1493 | 1490
Participants | 57 | 54

8. Secondary Outcome: Number of Participants Undergoing Renal-replacement Therapy
Time Frame: Indexed hospital stay
Measure: Count of Participants; unit: Participants
Arm/Group | Liberal Group | Restrictive Group
Number analyzed (Participants) | 1493 | 1490
Participants | 4 | 13

9. Secondary Outcome: Number of Participants With Pulmonary Edema
Time Frame: Indexed hospital stay
Measure: Count of Participants; unit: Participants
Arm/Group | Liberal Group | Restrictive Group
Number analyzed (Participants) | 1493 | 1490
Participants | 32 | 20

10. Secondary Outcome: Number of Participants With Unplanned Admission to ICU
Time Frame: 30 day
Measure: Count of Participants; unit: Participants
Arm/Group | Liberal Group | Restrictive Group
Number analyzed (Participants) | 1493 | 1490
Participants | 145 | 161

11. Secondary Outcome: Death
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Liberal Group | Restrictive Group
Number analyzed (Participants) | 1493 | 1490
Participants | 18 | 31

12. Secondary Outcome: Death
Time Frame: 12 month
Measure: Count of Participants; unit: Participants
Arm/Group | Liberal Group | Restrictive Group
Number analyzed (Participants) | 1493 | 1490
Participants | 96 | 95

ADVERSE EVENTS:
Arm/Group | Liberal Group | Restrictive Group
Serious Adverse Events (participants affected / at risk) | 103/1493 | 118/1490
Other Adverse Events (participants affected / at risk) | 205/1493 | 208/1490
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Liberal Group (N=1493) | Restrictive Group (N=1490)
Myocardial infarction (Cardiac disorders) | 23 | 13
Stroke (Vascular disorders) | 2 | 8
Other cardiovascular (Cardiac disorders) | 55 | 66
Thromboembolish (Vascular disorders) | 23 | 31
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Liberal Group (N=1493) | Restrictive Group (N=1490)
Other (Blood and lymphatic system disorders) | 205 | 208

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes